CLINICAL TRIAL: NCT02605044
Title: A Prospective, Multicenter, Randomized, Double Blind, Placebo-controlled, 2-parallel Groups, Phase 3 Study to Compare the Efficacy and Safety of Masitinib in Combination With FOLFIRI (Irinotecan, 5-fluorouracil and Folinic Acid) to Placebo in Combination With FOLFIRI in Second Line Treatment of Patients With Metastatic Colorectal Cancer
Brief Title: Masitinib in Combination With FOLFIRI for Second-line Treatment of Patients With Metastatic Colorectal Cancer
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Sponsor decision based on portfolio prioritization
Sponsor: AB Science (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AB12006
Record Dates: First submitted 2015-11-05; First posted 2015-11-16 (Estimated); Last update posted 2019-02-11 (Actual); Status verified 2019-02

CONDITIONS: Metastatic Colorectal Cancer
MeSH Terms: conditions — Colorectal Neoplasms | interventions — masitinib; IFL protocol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- Masitinib + FOLFIRI (Experimental): masitinib + FOLFIRI
  Interventions: Drug: Masitinib (AB1010); Drug: FOLFIRI
- Placebo + FOLFIRI (Placebo Comparator): Placebo + FOLFIRI
  Interventions: Drug: FOLFIRI

INTERVENTIONS:
Drug: Masitinib (AB1010)
  Arms: Masitinib + FOLFIRI
Drug: FOLFIRI

SUMMARY:
The objective is to compare the efficacy and safety of masitinib in combination with FOLFIRI ( irinotecan, 5-fluorouracil and folinic acid) to placebo in combination with FOLFIRI in second line treatment of patients.

ELIGIBILITY:
Inclusion Criteria:

* Patient with non-resectable metastatic colorectal cancer
* Metastatic disease not amenable to surgical resection
* Patient in second line treatment after progression according to RECIST criteria
* Patient with measurable lesions according to RECIST criteria (version 1.1)
* Patient eligible for a standard second line treatment with FOLFIRI
* Patient with ECOG ≤ 2
* Patient with adequate organ function
* Patient with life expectancy > 3 months
* Female or male patient ≥ 18
* Patient weight > 40 kg and BMI > 18

Exclusion Criteria:

* Patient who cannot receive FOLFIRI
* More than 1 prior chemotherapy regimens for metastatic colorectal cancer
* Pregnant, intent to be pregnant, or nursing female patient
* Patient with any chronic inflammatory bowel disease
* Patient treated for a cancer other than colorectal cancer within five years before enrollment
* Patient with an hepatic involvement > 50%
* Patient with active central nervous system (CNS) metastasis or history of CNS metastases
* Patient with an active infection
* Patient presenting with cardiac disorders
* Any previous treatment with an investigational agent or chemotherapy or biological agent within four weeks prior to baseline.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 123 (Actual)
Dates: Start 2014-01; Primary Completion 2017-12 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
Overall survival | From day of randomization to death, assessed for a maximum of 60 months
  Overall survival is defined as time in months from the randomization date to the date of death due to any cause. If a patient is not known to have died, then OS will be censored at the date of last known date patient alive.

SECONDARY OUTCOMES:
Survival rate | Every 24 weeks, assessed up to 60 months
  Survival rate is defined as the proportion of patients alive at each time point, estimated with Kaplan-Meier distribution
Progression Free Survival (PFS) | From day of randomization to disease progression or death, assessed for a maximum of 60 months
  Progression Free Survival is defined as the time from the randomization date until the date of earliest evidence of disease progression or death, for participants who progressed or died before subsequent cancer therapy. Disease progression will be assessed by the investigator on CT scan according to RECIST 1.1 criteria

CONTACTS AND LOCATIONS:
Overall Officials: Julien Taieb, PhD, MD, Principal Investigator — Hôpital Européen Georges Pompidou, Paris, France
Locations (3):
- Hopital Europeen George Pomipidou, Hepato-Gastro-enterologie, 20 rue Leblanc, Paris, France
- National Cancer Center, 11 Hospital Drive, Singapore, Singapore
- Hammersmith Hospital, Department of Cancer Medicine, Imperial College Healthcare Trust, Du Cane Road, London, United Kingdom